CLINICAL TRIAL: NCT06795022
Title: A Modular Phase I/II Open-label Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD9793, a T Cell-engaging Antibody Targeting Glypican-3 (GPC3) in Adult Participants With Advanced or Metastatic Solid Tumours (RHEA-1)
Brief Title: First in Human Study to Evaluate AZD9793 in Participants With Advanced or Metastatic Solid Tumours
Acronym: RHEA-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7040C00001
Record Dates: First submitted 2025-01-08; First posted 2025-01-27 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Glypican-3; GPC3; GPC3+ tumours; T cell-engaging antibody; TCE; AZD9793; Solid tumours; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Simpson-Golabi-Behmel syndrome

STUDY DESIGN:
Intervention Model Description: The study consists of individual modules each evaluating the safety and tolerability of AZD9793 dosed as monotherapy:
  Module 1: AZD9793 intravenous administration Module 2: AZD9793 subcutaneous administration
  Modules 1 and 2 each consist of two parts: Part A, Dose Escalation and Part B, Dose Expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1: AZD9793 Intravenous (IV) monotherapy (Experimental): Module 1: AZD9793 Intravenous (IV) monotherapy
  Interventions: Drug: AZD9793 Intravenous (IV) monotherapy
- Module 2: AZD9793 Subcutaneous (SC) monotherapy (Experimental): Module 2: AZD9793 Subcutaneous (SC) monotherapy
  Interventions: Drug: AZD9793 Subcutaneous (SC) monotherapy)

INTERVENTIONS:
Drug: AZD9793 Intravenous (IV) monotherapy — T cell-engaging antibody that targets GPC3 on tumour cells
  Arms: Module 1: AZD9793 Intravenous (IV) monotherapy
Drug: AZD9793 Subcutaneous (SC) monotherapy) — T cell-engaging antibody that targets GPC3 on tumour cells
  Arms: Module 2: AZD9793 Subcutaneous (SC) monotherapy

SUMMARY:
This research is designed to determine if experimental treatment with AZD9793, a T cell-engaging antibody that targets GPC3, is safe, tolerable and has anti-cancer activity in patients with advanced or metastatic solid tumours which are GPC3+.

DETAILED DESCRIPTION:
This is a first-time in human, modular Phase I/II, open-label multicentre study of AZD9793 monotherapy administered intravenously (Module 1), or AZD9793 monotherapy administered subcutaneously (Module 2) in patients with advanced or metastatic solid tumours. Each module contains dose-escalation (Part A) and dose-expansion (Part B).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 at the time of signing the informed consent.
* GPC3 positive tumour as determined by a central laboratory using an analytically validated IHC assay.
* Must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group Performance status (ECOG PS): 0-1 at screening.
* Predicted life expectancy of ≥ 12 weeks.
* Adequate organ and bone marrow function measured within 28 days prior to first dose as defined by the protocol.
* Contraceptive use by men or women should be consistent with local regulations, as defined by the protocol.
* Confirmed advanced recurrent and/or metastatic and/or unresectable HCC, which is histopathologically proven based on the criteria established by the World Health Organization.
* Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C.
* Child-Pugh Score class A.
* Previous therapy:

Part A: Patients who have received at least one prior line of standard systemic therapy for HCC as per National Comprehensive Cancer Network or other local scientific guidelines and for which a clinical study is the best option for next treatment based on prior response and/or tolerability and/or patient/investigator decision.

Part B: Patients must not have received more than one prior line of systemic therapy in the advanced recurrent and/or metastatic setting.

Key Exclusion Criteria:

* Unresolved toxicity from prior anticancer therapy, including imAEs, of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2 except for vitiligo, peripheral neuropathy related to prior anti-cancer therapy, alopecia, endocrine disorders that are controlled with replacement hormone therapy and asymptomatic laboratory abnormalities.
* Prior to enrolment, participation in another clinical study with an investigational product administered in the last 21 days or 5 half-lives whichever is shorter.
* CAR-T cell therapy within the last 6 months prior to enrolment on this study.
* Known allergy or hypersensitivity to AZD9793 or any of the excipients of the product as outlined in the IB.
* Requires chronic immunosuppressive therapy (including steroids > 10 mg prednisone/day or equivalent).
* Prior treatment with any therapy that is targeted to GPC3.
* Received radiation within 14 days prior to first dose of study treatment; palliative radiation to reduce the risk of tumour lysis syndrome (TLS) or CRS/neurotoxicity in participants with bulky disease is permitted.
* Undergone a major surgical procedure within 14 days prior to first dose of study treatment days to allow adequate healing
* Experienced unacceptable cytokine release syndrome (CRS) or Immune Effector Cell Associated Neurotoxicity (ICANS) following prior T cell engagers (TCE) or chimeric antigen receptor T (CAR-T) cell therapy.
* Previous history of hemophagocytic lymphohistiocytosis (HLH) / macrophage activation syndrome (MAS).
* Active or prior documented autoimmune or inflammatory disorders within 3 years of start of treatment.
* Cardiac conditions as defined by the protocol.
* History of thromboembolic event within the past 3 months prior to the scheduled first dose of study intervention.
* Central nervous system (CNS) metastases or CNS pathology, as defined by the protocol, within 3 months prior to consent.
* Infectious disease including active human immunodeficiency virus (HIV), and uncontrolled active systemic fungal, bacterial or other infection.
* Known fibrolamellar HCC, sarcomatoid HCC, or combined hepatocellular malignant cholangiocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-07-25 (Estimated)

PRIMARY OUTCOMES:
The number of patients with adverse events | From first dose of study drug up to 30 days post last dose and prior to start of subsequent anticancer therapy
  Number of patients with adverse events by system organ class and preferred term
The number of patients with serious adverse events | From first dose of study drug up to 30 days post last dose and prior to start of subsequent anticancer therapy
  Number of patients with serious adverse events by system organ class and preferred term
The number of patients with adverse events of special interest | From first dose of study drug up to 30 days post last dose and prior to start of subsequent anticancer therapy
  Number of patients with adverse events of special interest by system organ class and preferred term
The number of patients with dose-limiting toxicity (DLT), as defined in the protocol. | From date of first dose of study drug until the end of Cycle 1 (up to 28 days)
  Number of patients with at least 1 DLT. A DLT is a toxicity as defined in the protocol that occurs from the first dose of study drug up to and including the planned end of Cycle 1 (the DLT assessment period) that is assessed as unrelated to the disease or disease-related processes under investigation.
Objective Response Rate (ORR) [Dose expansion only] | From first dose of study drug to progressive disease or the last evaluable assessment in the absence of disease progression whichever comes first (up to approximately 2 years)
  The percentage of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST 1.1). Dose expansion only.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) [Dose escalation only] | From first dose of study drug to progressive disease or the last evaluable assessment in the absence of disease progression whichever comes first (up to approximately 2 years)
  The percentage of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST 1.1). Dose escalation only.
Best overall response (BOR) | From first dose until disease progression or the last evaluable assessment in the absence of progression (up to approximately 2 years)
  The best overall radiological visit response the participant achieves per RECIST 1.1 as assessed by the investigator.
Disease Control Rate (DCR) at 12 weeks | From first dose of study drug to progressive disease or last evaluable assessment in the absence of disease progression. [Expected to be measured for each patient at 12 weeks]
  Percentage of patients with confirmed complete or partial response or having stable disease maintained for >= 11 weeks, at 12 weeks from first dose, according to response criteria in solid tumours (RECIST 1.1).
Durable response rate (DRR) | From first documented objective response (subsequently confirmed) to the date of disease progression or the last evaluable assessment in the absence of progression (up to approximately 2 years)
  Percentage of participants who have a confirmed best overall response of CR or PR with a duration of at least 3 months, 6 months, 9 months, and 12 months.
Duration of response (DoR) | From the first documented objective response (subsequently confirmed) to progressive disease or death in absence of progression (up to approximately 2 years)
  The time from the date of first response until date of disease progression or death in the absence of disease progression, according to response criteria in solid tumours (RECIST 1.1).
Time To Response (TTR) | From start of study treatment until the date of first documented objective response, which is subsequently confirmed as assessed by the Investigator per RECIST 1.1 (up to approximately 2 years)
  The time from start of study treatment until the date of first documented objective response, which is subsequently confirmed as assessed by the Investigator per RECIST 1.1.
Progression free Survival (PFS) | From the start of study treatment to progressive disease or death due to any cause (up to approximately 2 years)
  The time from the start of study treatment until RECIST 1.1 defined disease progression or death in the absence of disease progression.
Overall Survival (OS) [Dose expansion only] | From the start of study treatment to death (up to approximately 2 years)
  The time from the start of study treatment until death due to any cause. Dose expansion only.
Pharmacokinetics of AZD9793: Maximum serum concentration of the study drug (Cmax) | From the first dose of study intervention, at predefined intervals throughout the study (up to approximately 2 years)
  Maximum observed serum concentration of the study drug
Pharmacokinetics of AZD9793: Area Under the concentration-time curve (AUC) | From the first dose of study intervention, at predefined intervals throughout the study (up to approximately 2 years)
  Area under the serum concentration-time curve
Pharmacokinetics of AZD9793: Clearance | From the first dose of study intervention, at predefined intervals throughout the study (up to approximately 2 years)
  A pharmacokinetic measurement of the volume of serum from which the study drug is completely removed per unit time.
Pharmacokinetics of AZD9793: Terminal elimination half-life (t 1/2) | From the first dose of study intervention, at predefined intervals throughout the study (up to approximately 2 years)
  Terminal elimination half life.
Immunogenicity of AZD9793 | From the first dose of study intervention, at predefined intervals throughout the study (up to approximately 2 years)
  The number and percentage of participants who develop anti-drug antibodies (ADAs) measured in serum
Change in CD8+ Levels | From time of Informed consent, at predefined intervals (including screening, on-treatment or end of treatment) throughout the study (up to approximately 2 years)
  Percentage change in CD8+ cells measured by IHC in samples taken pre and post treatment

CONTACTS AND LOCATIONS:
Locations (19):
- United States (6):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Houston, Texas
- China (4):
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Shanghai
- Hong Kong (2):
  - Research Site, Pokfulam
  - Research Site, Shatin
- Japan (2):
  - Research Site, Kashiwa
  - Research Site, Yokohama
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Pamplona
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/